CLINICAL TRIAL: NCT06590883
Title: The STatus Epilepticus Prognosis Study
Acronym: STEP
Status: Recruiting | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Teneille Gofton, Scientist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: REDA12409
Record Dates: First submitted 2024-07-16; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Status Epilepticus
Keywords: Neuroimaging; Neuronal injury; cognitive testing
MeSH Terms: conditions — Status Epilepticus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biospecimens include blood and CSF
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to improve the prognosis of patients who present with Status Epilepticus (SE). In the first part of this study, the investigators aim to find better markers of good and poor outcomes of SE patients while in the ICU. The objective is to measure the levels of brain protein micro-particles that are detectable in blood samples. The investigators seek to determine whether elevated levels of micro-particles in the bloodstream in SE patients can be used to predict the eventual outcome of survivors. The goal of the second part of the study is to evaluate long-term cognitive outcomes in survivors of SE To date, there is no reliable information to inform what cognitive recovery is like for survivors of SE after ICU discharge. The objective is to use the Creyos cognitive testing platform to assess different domains of cognitive function for up to 1 year after SE onset. Patients who have pre-existing epilepsy but have not had status epilepticus will serve as patient controls for the cognitive testing portion of this study. The third part of this study will evaluate brain changes in survivors of refractory SE. To date, there are no known studies that document to what extent the anatomy of the brain changes following SE. The objective is to characterize these changes by conducting two brain research scans 6 months apart. Patients will be invited to Robart's Research Institute for a scan 1-3 months and 6-8 months (6 months apart) after refractory SE to measure structural and functional changes in the brain throughout the recovery process.

DETAILED DESCRIPTION:
Treatment guidelines and predictive markers of neurologic recovery in status epilepticus (SE) and refractory SE are inadequate, which makes prognostication of neurological outcome a substantial clinical challenge. Given that SE is the second most common neurological emergency, there is an urgent need for novel biomarkers to predict outcome of patients admitted in the ICU. Given this limited data, evidence of CNS injury and inflammation may serve as biomarkers of SE severity and prognosis.

The etiology of seizures, patient age and extent of epileptiform activity are thought to be related to long neurocognitive impairments in survivors of SE/RSE. However, measures of outcome are often dichotomized as "good" and "poor", and the extent of cognitive dysfunction and the specific cognitive processes that are impaired stand to be elucidated. Additionally, the literature characterizing cognitive function after SE is heterogenous, with variability in the assessment tools and time points for neurocognitive function which leads to limited understanding of the true incidence, severity, and long-term implications of cognitive impairment.

In recent years, there has been an expansion of available cognitive assessment tools that can be self-administered remotely, overcoming the previous barriers to patient assessment. One such tool is the Creyos platform, a web-based neurocognitive battery consisting of 12 cognitive tasks (designed as online games) assessing cognitive function across various domains, including concentration, memory, verbal skills, and reasoning. The Creyos tests have the advantage of allowing for remote self-administration, which means that patients from a broader geographic area can complete outcome measures without having to travel for assessment. Including more patients in this way will undoubtedly improve research generalizability. In a recent pilot study, the Creyos battery was used in a cohort of ICU patients and showed that it is both feasible and able to identify cognitive impairment in several domains. These results demonstrate that web-based studies of cognition are not only possible but provide a novel opportunity for evaluating neurocognitive impairments in an accessible manner that would not be feasible using traditional methods.

Persistent epileptiform activity is thought to contribute to neuronal death following RSE ultimately resulting in progressive brain atrophy. Previous literature suggests that duration of anesthetic therapy and length of hospital stay are related to loss of parenchymal volume, and hippocampal and diffuse cerebral atrophy on MRI are more likely to be associated with worse functional outcomes. In people with epilepsy, neuroimaging techniques such as volumetric analysis of the hippocampus and associated cortices have shown evidence of volumetric changes that are predictive of reduced cognitive abilities. However, the vast majority of the current literature consists of retrospective analyses, and there are no known studies that have directly assessed the relationship between cerebral damage following RSE and functional/cognitive outcomes.

Functional and diffusion tensor imaging (fMRI/DTI) are two sophisticated neuroimaging methods that can be used to accurately measure the functional and structural integrity of the brain, respectively, with high precision and accuracy. These methods have been used in the past to image people with epilepsy, and several studies have shown large-scale functional network reorganization in this patient group (for review, see Gonen, 2020). Interestingly, correlations to disease duration and severity (e.g., drug resistance) have also been found in these studies. Characterizing functional and structural changes in survivors of RSE provides a unique opportunity for investigating the anatomical and functional correlates that may underlie impaired cognition and reduced quality of life, and will likely lead to an in-depth understanding of how acute epileptiform activity can alter the structural and functional mechanics of the brain.

The overall goal of this study is to comprehensively evaluate the acute and long-term effects of Status Epilepticus on the brain. The overarching research question is: do acute markers of neural degeneration that can be detected in blood plasma predict the long-term outcome of patients with Status Epilepticus? And, do these markers relate to cognitive and functional outcomes? The investigators hypothesize that patients who have higher levels of markers of neuronal degeneration in their blood samples from the ICU will have poor clinical outcomes, as indexed by their scores on the Creyos cognitive battery. The investigators also hypothesize that refractory status patients who have higher levels of markers of neuronal degeneration in their bloodstream in the ICU will have greater structural and functional alterations in their brain at ~1 and ~6 months post-seizure onset.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years of age
* SE requiring admission to critical care
* Developed SE while in ICU
* No history of a neurologic condition, other than epilepsy, that would impact cognition (Dementia, Parkinson's disease, Alzheimer's disease)
* Absence of devastating neurologic injury (cardiac arrest, stroke, traumatic brain injury)

In addition, for non-SE epilepsy controls for Creyos task:

* People with epilepsy
* No history of status epilepticus
* Patient has not stereotaxic EEG monitoring
* English speaking
* No history of a neurologic condition, other than epilepsy, that would impact cognition (Dementia, Parkinson's disease, Alzheimer's disease)

In addition, for follow up MRI purposes only:

* Diagnosed with refractory status epilepticus while in ICU
* No MRI contraindications (metal in body, pacemakers, etc.)

Inclusion Criteria Healthy Control Population for MRI imaging:

* No history of a neurologic condition that would impact cognition (Dementia, Parkinson's disease, Alzheimer's disease)
* No MRI contraindications (metal in body, pacemakers, etc.)

Exclusion Criteria:

* patients not meeting inclusion criteria
* acute brain injury or brain tumour as immediate cause of status epilepticus

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Overall, 50 status epilepticus patients will be identified in three ICUs in London, Ontario over three years. Study participants will be SE patients admitted to either the medical-surgical intensive care unit (MSICU), the cardiac surgery recovery unit (CSRU) or the critical care trauma centre (CCTC) at London Health Sciences Centre. Up to 50 people with epilepsy will also be recruited from the Neurology outpatient clinic and Epilepsy Monitoring Unit at University Hospital to serve as patient controls for the neurocognitive testing component of this study. The investigators expect up to 12 Refractory Status Patients to be recruited for objective 3 and an equivalent number of healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-11-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
serum extracellular microvesicle analysis | Day 1-21 after admission
  analysis of blood samples to assess for markers of neuronal injury
Creyos cognitive battery | 1-12 months after admission
  Longitudinal online cognitive assessment
functional MRI | 3-6 months after admission
  Longitudinal assessment in patients with refractory status epilepticus

SECONDARY OUTCOMES:
Function outcome | 1-12 months after admission
  modified Rankin Scale - Scores from 0-6 with lower scores indicating a better outcome (0=no symptoms; 6=death)
Function outcome | 1-12 months after admission
  Telephone Interview for Cognitive Status - maximum 41 points, minimum 0 points, higher scores indicate better outcome
Function outcome | 1-12 months after admission
  Neuro-Quality of Life - Scores 0.5 - 1.0 SD worse than the mean = mild symptoms/impairment; Scores 1.0 - 2.0 SD worse than the mean = moderate symptoms/impairment; Scores 2.0 SD or more worse than the mean = severe symptoms/impairment

CONTACTS AND LOCATIONS:
Locations (1):
- Lawson Health Research Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Requests for access to data will be considered on an individual basis with approval of the Western Health Sciences Research Ethics Board. The informed consent does not include open sharing of the data.